CLINICAL TRIAL: NCT04772586
Title: Sarcopenia and Mechanical Ventilation in Older Patient Admitted With COVID-19 Infection
Brief Title: Sarcopenia and Mechanical Ventilation in Older Patients Admitted Due to COVID-19
Acronym: SARCO-V
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Murielle Surquin, Prof Dr Murielle Surquin MD PhD, Brugmann University Hospital
Other Study IDs: SARCO-V_2020/110
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Mechanical ventilation; Older patients; COVID-19
MeSH Terms: conditions — Sarcopenia; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SarcoV study aims at assessing the association between sarcopenia and the indication of mechanical ventilation in older hospitalized patients due to COVID-19 infection

DETAILED DESCRIPTION:
Sarcopenia is disease associated with poor clinical outcomes. In critical ill chirurgical patients, sarcopenia is associated with difficult to wean of mechanical ventilation. The association between sarcopenia and mechanical ventilation is poorly studied in medical patients. COVID-19 pandemic has led a lot of medical patient to be admitted in intensive care units due to acute respiratory failure with need of mechanical ventilation support.

The primary objective is to determine if sarcopenia in critically-ill older patients with COVID-19 is associated with the indication of mechanical ventilation. Secondarily, the study aims at determining if sarcopenia is associated with difficult to wean and mortality in critically-ill older patients with COVID-19.

ELIGIBILITY:
Inclusion criteria

* Consecutive patients aged 60 and older
* Admission in an acute care unit in Brugmann university hospital due to a COVID-19 possible or confirmed infection. A infection was considered confirmed in presence of a positive molecular test by Polymerase-chain reaction (PCR), following the Belgian Public Health Department recommendations (Sciensano recommendations).

Exclusion criteria

* Patients unable to perform a grip-strength measurement due to any rheumatological or neurological condition.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 60 and older admitted in an acute care unit of Brugmann university hospital due to COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Indication of mechanical ventilation | Through study completion, an average of 60 days
  Association between probable sarcopenia and the indication of mechanical ventilation in patients with COVID-19 infection.
  Mechanical ventilation was considered by non-invasive ventilation or invasive ventilation. For purpose of analysis, it was defined as a binary outcome (yes(no).
  Probable sarcopenia probable was defined according to the revised European consensus on definition and diagnosis of sarcopenia (EWGSOP2). For purpose of analysis, it was defined as a binary condition (yes/no).

SECONDARY OUTCOMES:
Evaluate difficult-to-wean in mechanical ventilation | Through study completion, an average of 60 days
  Difficult to wean in mechanical ventilation is defined if the patient required more than 7 days of mechanical ventilation from the first spontaneous breath test or if the patient was reintubated within 48 hours after extubation. For purpose of analysis, it was considered as a binary outcome (yes/no)
All-cause mortality | Through study completion, an average of 60 days
  Vital status during hospital admission, at 30- and 60-day follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Brugmann university hospital, Brussels, Belgium

REFERENCES:
- [Background] Kou HW, Yeh CH, Tsai HI, Hsu CC, Hsieh YC, Chen WT, Cheng HT, Yu MC, Lee CW. Sarcopenia is an effective predictor of difficult-to-wean and mortality among critically ill surgical patients. PLoS One. 2019 Aug 8;14(8):e0220699. doi: 10.1371/journal.pone.0220699. eCollection 2019. PMID 31393937
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- See also: Definition of a confirmed COVID-19 case and National recommendations for the request of PCR test for COVID-19 in Belgium by the Belgian Public Health Department (Sciensano) — https://covid-19.sciensano.be/fr/covid-19-definition-de-cas-et-testing